CLINICAL TRIAL: NCT02953444
Title: The Feasibility and Efficacy of an Extremely Brief Mindfulness Practice
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient personnel to complete the study.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00072981
Record Dates: First submitted 2016-11-01; First posted 2016-11-02 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Depression; Anxiety; Mental Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wait List Control (No Intervention): Participants receive daily email surveys for two weeks before being given access to the brief-mindfulness-practice training materials.
- Thirty-Second Mindfulness Practice (Experimental): Participants watch a ten minute mindfulness training video then are given electronic access to an audio recording of guidance for a thirty-second mindfulness meditation practice. Participants are asked to complete this practice using the audio-recorded guidance at least three times a day for two weeks. Participants are sent daily emails that include reminders to complete the practice and a link to a brief online survey.
  Interventions: Other: Thirty-Second Mindfulness Practice
- Three-Minute Mindfulness Practice (Active Comparator): Participants watch a ten minute mindfulness training video then are given electronic access to an audio recording of guidance for a three minute mindfulness meditation practice. Participants are asked to complete this practice using the audio-recorded guidance at least three times a day for two weeks. Participants are sent daily emails that include reminders to complete the practice and a link to a brief online survey.
  Interventions: Other: Three-Minute Mindfulness Practice

INTERVENTIONS:
Other: Thirty-Second Mindfulness Practice
  Arms: Thirty-Second Mindfulness Practice
Other: Three-Minute Mindfulness Practice
  Arms: Three-Minute Mindfulness Practice

SUMMARY:
This study will assess the efficacy of brief mindfulness practices on improving mental health in adults who are currently in treatment for mental health concerns. From online instructional videos, each participant will learn a thirty-second or three-minute mindfulness practice that is to be performed at least three times daily over two weeks.

DETAILED DESCRIPTION:
Mindfulness meditation and mindfulness-based therapies have been shown to improve many aspects of psychological functioning in individuals with mental health problems.

The purpose of this study is to assess the feasibility, acceptability, and efficacy in improving mental health of brief mindfulness practices in adults currently in treatment for mental health concerns. The entire study will be administered online. From online instructional videos, each participant will learn a thirty-second or three-minute mindfulness practice that is to be performed at least three times daily over two weeks. A delayed-treatment control group will begin the intervention after a two-week waiting period.

ELIGIBILITY:
Inclusion Criteria:

* Regular internet access
* Able to listen to audio files
* Currently receiving outpatient care
* No change in type of psychotherapy during the past month
* If taking medications, a stable, unchanging prescription for the previous month
* Willingness to sign release of mental health care information
* Capacity to provide informed consent

Exclusion Criteria:

* Does not speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-11; Primary Completion 2018-09-09 (Actual); Study Completion 2018-09-09 (Actual)

PRIMARY OUTCOMES:
Change in trait mindfulness as measured by the Five Facet Mindfulness Questionnaire (Baer et al. 2006) | Baseline, 2 weeks and 4 weeks
Change in perceived stress as measured by the Perceived Stress Scale (Cohen, Kamarck, & Mermelstein, 1983) | Baseline, 2 weeks and 4 weeks
Change in anxiety symptoms as measured by the GAD-7, Generalized Anxiety Disorder Scale (Spitzer, Kroenke, Williams, & Löwe, 2006) | Baseline, 2 weeks and 4 weeks
Change in mood as measured by the Positive and Negative Affect Schedule (Watson, Clark, & Tellegen, 1988) | Baseline, 2 weeks and 4 weeks
Change in quality of life as measured by the Medical Outcomes Study 36-Item Short-Form Health Survey (Ware & Sherbourne, 1992) | Baseline, 2 weeks and 4 weeks
Change in depression symptoms as measured by the PHQ-8, Patient Health Questionnaire - depression module (Spitzer, Kroenke, & Williams, 1999) | Baseline, 2 weeks and 4 weeks

SECONDARY OUTCOMES:
Group difference in intervention's acceptability as measured by qualitative questions | 1 week into intervention
Group difference in adherence as measured by frequency of daily brief mindfulness practice use | Daily for two weeks of intervention
Group difference in continued brief mindfulness practice use as measured by follow-up question | Follow up (two weeks after intervention)
Change in daily mood measured on a visual analogue scale | Daily for two weeks of intervention
Change in daily stress level measured on a visual analogue scale | Daily for two weeks of intervention
Change in empathy as measured by the Interpersonal Reactivity Index (Davis, 1980) and four questions adapted from Hawk, Fischer and Van Kleef, (2011) | Baseline, 2 weeks and 4 weeks
Change in perspective taking as measured by questions adapted from Hawk, Fischer and Van Kleef, (2011) | Baseline, 2 weeks and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Moria Smoski, Ph.D, Principal Investigator — Duke University
Locations (1):
- Duke Office of Clinical Research REDCap Online Data Collection Software, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Khoury B, Lecomte T, Fortin G, Masse M, Therien P, Bouchard V, Chapleau MA, Paquin K, Hofmann SG. Mindfulness-based therapy: a comprehensive meta-analysis. Clin Psychol Rev. 2013 Aug;33(6):763-71. doi: 10.1016/j.cpr.2013.05.005. Epub 2013 Jun 7. PMID 23796855
- [Background] Davis, M.H. (1980). A multidimensional approach to individual differences in empathy. Catalogue of Selected Documents in Psychology, 10, MS. 2124, p. 85.
- [Background] Hawk ST, Fischer AH, Van Kleef GA. Taking your place or matching your face: two paths to empathic embarrassment. Emotion. 2011 Jun;11(3):502-13. doi: 10.1037/a0022762. PMID 21668103